CLINICAL TRIAL: NCT01736098
Title: Evaluation of Energy Balance at High vs. Low Energy Flux - Energy Flux Study
Brief Title: The Energy Flux Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: The Coca-Cola Company (Industry)
Responsible Party: Principal Investigator, Sarah Schumacher, Director, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00018017
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Energy Flux (Experimental): Energy Flux Exercise Intervention: 7kcal/kg/day at 5 days/week of energy expenditure and matching energy intake
  Interventions: Other: Energy Flux Exercise Intervention
- Medium Energy Flux (Experimental): Energy Flux Exercise Intervention: 3.5kcal/kg/day at 5 days/week of energy expenditure and matching energy intake
  Interventions: Other: Energy Flux Exercise Intervention
- Low Energy Flux (No Intervention): No Intervention: maintain normal lifestyle

INTERVENTIONS:
Other: Energy Flux Exercise Intervention — Comparison of high, medium and low energy flux groups with all groups matching energy intake and expenditure
  Arms: High Energy Flux; Medium Energy Flux

SUMMARY:
The focus of this randomized clinical trial study is an examination of the effects of maintaining energy balance at different energy fluxes. It will address the primary question: Are there increased health benefits related to body composition and metabolic function associated with maintaining energy balance at a high energy flux as compared to a low energy flux?

DETAILED DESCRIPTION:
We will randomly assign 75 sedentary but healthy individuals to one of two exercise groups or a non-exercise group. We will follow the individuals for 6 months during the intervention period. Both groups will maintain weight by matching energy intake and expenditure (thus the exercise group will consume more calories).

ELIGIBILITY:
Inclusion Criteria:

* BMI <35
* 21-45 years of age
* Fasting plasma glucose <126 mg/dl
* Current medications must have been prescribed for 3 or more months and stable
* Internet access
* Able to participate in a somewhat strenuous physical exercise program
* Able to provide informed consent for participation in a research study

Exclusion Criteria:

* Currently participating in a weight loss or exercise intervention / program
* Planning to have weight loss surgery
* Weight change >5 lb in last 12 months
* Currently taking any of the following: hormone replacement therapy, beta blockers, allergy shots or systematic corticosteroids (except inhalers)
* Significant cardiovascular disease or disorders including but not limited to: serious arrhythmias, cardiomyopathy, congestive heart failure, stroke or transient ischemic cerebral attacks, peripheral vascular disease with intermittent claudication, acute, chronic or recurrent thrombophlebitis, Stage II or Stage III hypertension, myocardial infarction or abnormal exercise stress test.
* Medical history with presence of significant conditions or disease that may interfere with study, recent surgery
* Pregnant or actively trying to become pregnant
* Gave birth in the last 12 months or <6 months post-lactation
* > 90th percentile on the Brief Symptom Inventory [BSI]
* Planning to move from the area in the next 8 months
* Other medical, psychiatric or behavioral factors that in the judgment of the principal investigator may interfere with study participation or the ability ot follow the intervention protocol. Upon identification of individuals with suicidal ideation or other dangerous conditions, the individual will be contacted and told to immediately go to a medical emergency room.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in anthropometrics | From baseline to 6 months
  Changes in lean and fat mass

OTHER OUTCOMES:
Changes in blood lipids | Baseline to 6 months
  Change in serum triglycerides
Changes in blood lipids | Baseline to 6 months
  Change in High Density Lipoprotein [HDL]
Changes in blood lipids | Baseline to 6 months
  Change in Low Density Lipoprotein [LDL]
Changes in blood lipids | Baseline to 6 months
  Change in LDL particle size
Change in functional measurements | Baseline to 6 months
  Change in cardiorespiratory fitness through graded exercise testing
Change in functional measurements | Baseline to 6 months
  Change in resting metabolic rate
Changes in markers of systemic inflammation | Baseline to 6 months
  Change in tumor necrosis factor-alpha [TNF-alpha]
Changes in markers of systemic inflammation | Baseline to 6 months
  Change in C reactive protein [CRP]
Changes in markers of systemic inflammation | Baseline to 6 months
  Change in interleukin-6 [IL-6]
Changes in triglyceride / cholesterol transport | Baseline to 6 months
  Change in Apolipoprotein E [ApoE]
Changes in triglyceride / cholesterol transport | Baseline to 6 months
  Change in Apolipoprotein B-48 [ApoB-48]
Changes in triglyceride / cholesterol transport | Baseline to 6 months
  Change in Apolipoprotein B-100 [ApoB-100]
Change in the index of fatty acid metabolism | Baseline to 6 months
  Change in serum 3 hydroxybutyric acid
Changes in carbohydrate metabolism | Baseline to 6 months
  Change in serum insulin
Changes in carbohydrate metabolism | Baseline to 6 months
  Change in glucose
Changes in carbohydrate metabolism | Baseline to 6 months
  Change in hemoglobin A1c [HbA1c]
Changes in energy intake | From Baseline to 6 months
Changes in energy expenditure | From Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hand, Ph.D, Principal Investigator — University of South Carolina; Steven Blair, Ph.D, Principal Investigator — University of South Carolina
Locations (1):
- Public Health Research Center, University of South Carolina, Columbia, South Carolina, United States